CLINICAL TRIAL: NCT02296216
Title: LateR-Ac Study: Late Effects of Radiosurgery on Acromegaly Study
Brief Title: Late Effects of Radiosurgery on Acromegaly Study
Acronym: LateRAc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-08; RCAPHM14_0079 (Registry Identifier: APHM)
Record Dates: First submitted 2014-10-28; First posted 2014-11-20 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acromegaly
Keywords: have been treated or not treated by Gamma Knife Radiosurgery
MeSH Terms: conditions — Acromegaly | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed patients (Active Comparator): Exposed patients have been treated by Gamma Knife Radiosurgery after unsuccessful surgery 10-20 years before inclusion
  Interventions: Device: Gamma Knife radiosurgery
- Unexposed patients (Placebo Comparator): Unexposed patients have not been treated by Gamma Knife Radiosurgery after unsuccessful surgery 10-20 years before inclusion
  Interventions: Device: Gamma Knife radiosurgery

INTERVENTIONS:
Device: Gamma Knife radiosurgery — To determine potential long-term (superior to 10 years) extra-pituitary side-effects of Gamma Knife radiosurgery in patients treated for Acromegaly

SUMMARY:
Transsphenoidal surgery is the first-line treatment of acromegaly. Adjunctive radiotherapy can be necessary when surgery is ineffective to avoid a prolonged medical treatment. Several studies reported long-term extra-pituitary side-effects of conventional radiotherapy. However, none has evaluated potential side-effects induced by Gamma Knife radiosurgery, a highly precise stereotactic technique, that has been used as an effective treatment of acromegaly.

Aims of the study: To determine potential long-term (superior to 10 years) extra-pituitary side-effects of Gamma Knife radiosurgery in patients treated for Acromegaly.

Methods: Transversal exposed/unexposed study. Exposed patients have been treated by Gamma Knife Radiosurgery after unsuccessful surgery 10-20 years before inclusion, whereas unexposed patients have been treated by somatostatin analogs after unsuccessful surgery for at least 10 years before inclusion. 80 Patients (40 patients/group) will be evaluated in terms of cognitive dysfunction, quality of life, secondary tumor, stroke, pituitary deficits and growth hormone control of hypersecretion. Recruitment is planned to last for 2 years.

Expected results: We should be able to determine whether Gamma Knife radiosurgery is a long-term safe technique. This result might modify the management and follow-up of patients with acromegaly unsuccessfully treated by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject, man or woman, whose age is greater than or equal to 18 years;
* Subject has a combination of defined values plus Insulin Like Growth Factor-1 and no braking growth hormone (<1.2 milli-International unit/L) during an oral glucose tolerance acromegaly.
* Exposed: Subject with a surgically treated in remission with or without drug treatment somatostatinergic, acromegaly who received treatment with Gamma Knife radiosurgery within not less than 10 years and less than or equal to 20 years.
* Not exposed: Subject with a surgically treated acromegaly controlled by treatment somatostatinergic, not having received Gamma Knife radiosurgery.
* Subjects with thyroid under standardized assessment Levothyrox® inclusion in case of deficit associated thyroid stimulating;
* Topic supported in a project partner services;
* Subjects who have signed a written informed consent and agreeing to abide by the instructions of the protocol.

Exclusion Criteria:

* Minor or over the age of 75 years subject,
* Subjects with acromegaly resistant to somatostatinergic, or that required power is pegvisomant or cabergoline
* Subjects who received two pituitary neurosurgical treatment or treatment with conventional radiotherapy or radiosurgery treatments 2
* Pregnant or lactating woman,
* Topic is not affiliated with the social security system, or private about freedom;
* Subject refusing to participate in the study or not signing the informed consent;
* Subject with malignant disease known evolutionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
The cognitive assessment measure a subject as cognitively preserved or cognitively impaired | 24 months
  Assessment of cognitive functions based on:
  * Evaluation of the memory component : Test Grober and Buschke.
  * Cognitive functions : Tests Stroop and Trail making test.
  * Evaluation of the care component and concentration : Paced Auditory Serial Addition Test.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France